CLINICAL TRIAL: NCT05561660
Title: Comparison of the Effect of Device Closure in Alleviating Migraine With Patent Foramen Oval (COMPETE-2)
Brief Title: COMParison of the EffecT of dEvice Closure in Alleviating Migraine With PFO (COMPETE-2)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Project Manager, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-1748
Record Dates: First submitted 2022-09-28; First posted 2022-09-30 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Migraine; Patent Foramen Ovale
MeSH Terms: conditions — Migraine Disorders; Foramen Ovale, Patent | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PFO closure (Experimental)
  Interventions: Device: PFO device closure
- Shame procedure (Sham Comparator)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Device: PFO device closure — Participants randomized into this group will take PFO device closure.
  Arms: PFO closure
Drug: Aspirin — Participants randomized into this group will take aspirin 200mg qd for 6 months.
  Arms: Shame procedure

SUMMARY:
Migraine attacks are episodic disorder that affects approximately 12% of the population, and studies have shown that 41-48% of migraineurs have a combination of patent foramen ovale (PFO). Clinical Observational studies have been linking PFO occlusion with the effectiveness in improving migraine symptoms and reducing the frequency of attacks. However, several RCTs have shown negative primary results, making it unclear whether PFO occlusion is effective in treating migraine. Our study is a prospective, double-blind, multi-center, and randomized study designed to test the effectiveness of migraine alleviation by performing percutaneous closure of patent foramen ovale in patients who are also diagnosed with PFO and migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 ；
2. Diagnosed migraine by ICHD-3
3. History of migraine longer than 1 year
4. TCD/TTE/TEE diagnosed patent foramen ovale
5. Willing to participant and agree to follow-ups
6. Undertook medication therapy for three months without a responder rate higher or equal to 50%

Exclusion Criteria:

1. Migraine caused by other reason
2. Had TIA/stroke history
3. Hypersensitive or hyposensitive to the study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Responder rate | From baseline period to 12-month treatment period
  Defined as a 50% reduction from the monthly number of migraine attacks during the baseline phase to the monthly number of migraine attacks during the treatment phase.
Treatment safety | From baseline period to 12-month treatment period
  Adverse events after medication treatment
  Adverse events after medication treatment
  Adverse events after medication treatment
  Adverse events after medication treatment
  Adverse events after medication treatment

SECONDARY OUTCOMES:
Migraine days change per month | From baseline period to 12-month treatment period
  Change in the mean number of migraine days from baseline to treatment phase.
Number of migraine attacks change per month | From baseline period to 12-month treatment period
  Change in the mean number of migraine attacks from baseline to treatment phase.
Percentage of migraine change | From baseline period to 12-month treatment period
  Participants experienced 75%, or greater reduction in migraine headache attacks during treatment phase as compared to baseline phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China